CLINICAL TRIAL: NCT05263245
Title: The Pharmacological Effects of Using Cabozantinib With a Light Breakfast: the Skippy 1 Study
Brief Title: The Pharmacological Effects of Using Cabozantinib With a Light Breakfast
Acronym: Skippy 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: dr. Tom van der Hulle (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, dr. Tom van der Hulle, Principal Investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 81846
Record Dates: First submitted 2022-02-11; First posted 2022-03-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Carcinoma, Renal Cell / drug therapy; Cabozantinib; Angiogenesis Inhibitors / pharmacokinetics; Food-drug interactions
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma

STUDY DESIGN:
Intervention Model Description: Multicenter open label randomized cross-over design. Patients will be randomized to start with the experimental or standard regimen. In the experimental regimen, patients will take cabozantinib with a light breakfast. In the standard regimen, patients will take cabozantinib in fasted state. After all pharmacokinetic samples have been completed, patients will switch to the other regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard regimen (No Intervention): Patients will continue to use cabozantinib in fasted state, as part of standard of care, in the recommended dose as prior to enrollment in the study.
- Experimental regimen (Experimental): Patients will take the prior recommended dose cabozantinib with a light breakfast.
  Interventions: Other: Light breakfast

INTERVENTIONS:
Other: Light breakfast — Light breakfast, standardized by 7 menu options for patients. All breakfast options contain the same amount of fat (9-10 g). Example of a menu: 150 ml full-fat yoghurt, 40 gram muesli with sugar, 1 glass of tea.
  Arms: Experimental regimen

SUMMARY:
Cabozantinib is a drug which is used to treat metastasized kidney cancer. While it works well, it has a lot of side effects and is quite expensive (€213,- every tablet, €6403,- every month). The standard recommended dose is 60 mg once a day, taken in fasted state. This means patients are not allowed to eat at least 2 hours before and one hour after taking cabozantinib. In daily practice, this is difficult for patients. It might be that by taking with breakfast the chance of side effects like nausea and diarrhea decreases. If patients take cabozantinib with breakfast, the body will have a higher uptake of the drug.

Often the dose of cabozantinib has to be lowered due to side effects. All tablets cabozantinib have the same price, despite how many milligrams are in the tablets. Cabozantinib stays in the body for a long time after ingestion. It takes approximately 120 hours before half of the medicine has left the body. This means it might not be necessary to take cabozantinib every day. Therefore, it is interesting to investigate if taking cabozantinib with breakfast makes it possible to skip taking cabozantinib once in a while. In this study, the investigators want to investigate to what extent the exposure of cabozantinib increases after ingestion with a light breakfast. The results from this study will be used for the development of alternative dosing regimens with cabozantinib tablets of 60 mg taken with a light breakfast including skipping days.

In this study, patients will randomized to start with taking cabozantinib in fasted state (standard regimen) and taking cabozantinib with a light breakfast (experimental regimen). Menu options will be provided. After at least 4 weeks taking cabozantinib according to the randomized regimen, patients will be submitted to the hospital for one day to measure the amount of cabozantinib in the blood at several points of time. This will be measured by venepuncture and fingerprick microsampling. When all blood samples have been collected, the patient will switch to the other regimen. After at least 4 weeks taking cabozantinib according to the second regimen, venous blood samples will be collected in exactly the same way. After all patients have completed the study, an analysis will be performed to determine the change in exposure to cabozantinib when it is taken with a light breakfast. The results will be used in order to determine the definitive experimental dosing regimens that will be investigated a subsequent study. Patients will be monitored for side effects, especially nausea and/or diarrhea.

The primary goal is to investigate to what extent the exposure of cabozantinib increases by taking cabozantinib with a light breakfast compared to taking cabozantinib in fasted state. The secondary objective is to investigate the analytical feasibility of microsampling (finger prick) for cabozantinib concentration measurements and to monitor side effects.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Aged 18 years or older;
* Histologically confirmed advanced renal cell carcinoma;
* Receiving cabozantinib as monotherapy as treatment for RCC;
* At least 4 weeks on a stable dosage of cabozantinib;
* Acceptable tolerability and the need for dose reductions or treatment interruptions has been estimated as low;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Estimated life expectancy of ≥ 6 months;
* No response evaluation planned during the study period;
* Cabozantinib trough concentration ≤1125 ng/ml in steady state

Exclusion Criteria:

* Inability to follow the recommended light breakfast;
* Gastro-intestinal abnormalities influencing the absorption of cabozantinib, including active inflammatory bowel diseases, malabsorption syndrome and prior major surgery of the stomach, pancreas, liver or smaller bowel.
* Use of moderate or strong inhibitor of cytochrome P450 enzymes within 1 month of start of treatment with cabozantinib, including ketoconazole, grape fruit juice, clarithromycin, erythromycin, itraconazole and ritonavir.
* Use of moderate or strong inducer of cytochrome P450 enzymes within 1 month of start of treatment with cabozantinib, including rifampicin, phenytoin, carbamazepine, phenobarbital and herbal preparations containing St. John's Wort.
* Use of inhibitor of multidrug resistance-associated protein 2 within 1 month of start of treatment with cabozantinib, including cyclosporine, delavirdine, efavirenz, emtricitabine, benzbromarone and probenecid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) | At both hospital admissions after at least 28 days on the regimen (t = 0, 1, 2, 3, 4, 5, 6, 8 and 24 hours)
  Increase of the area under the concentration-time curve (AUC) of the experimental regimen compared to the standard regimen

SECONDARY OUTCOMES:
Analytical feasibility | At both hospital admissions after at least 28 days on the regimen (t = 0, 1, 2, 3, 4)
  Analytical correlation/agreement between venapuncture (plasma) measurements and microsampling (whole blood and capillary plasma) measurements
Adverse events | At inclusion and at both hospital admissions after at least 28 days on the regimen
  The total number of patients experiencing (S)AEs

CONTACTS AND LOCATIONS:
Overall Officials: Tom van der Hulle, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided
To be determined in detail

REFERENCES:
- [Derived] Rieborn A, Guchelaar NAD, van Gelder T, Gelderblom H, Luelmo SAC, Kerssemakers N, Hamberg PAP, Koolen SLW, Mathijssen RHJ, Moes DJAR, van der Hulle T. The Effect of Taking Cabozantinib with a Light Breakfast: A Randomized Crossover Pharmacokinetic Study (SKIPPY 1). Clin Pharmacokinet. 2026 Jan 19. doi: 10.1007/s40262-025-01612-2. Online ahead of print. PMID 41555108